CLINICAL TRIAL: NCT02879019
Title: 12 Weeks of Walking Exercise Training in Women With Peripheral Artery Disease: A Sub-study of GrEnADa-project
Brief Title: Walking Training in Peripheral Artery Disease (GrEnADa Sub-study)
Acronym: GrEnADa
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not started due to lack of funding
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Véronique Cornelissen, PhD, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 150716_GrenSub
Record Dates: First submitted 2016-08-11; First posted 2016-08-25 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Peripheral Artery Disease; Intermittent Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stretching exercise group (Sham Comparator): Patients will receive two session per week of stretching classes.
  Interventions: Other: Stretching exercise group
- Walking training group (Experimental): Patients will perform two walking sessions per week.
  Interventions: Other: Walking training group

INTERVENTIONS:
Other: Stretching exercise group — In each stretching class, approximately 20 exercises will be performed. The total duration of the session will be approximately 30 minutes.
  Arms: Stretching exercise group
Other: Walking training group — Patients will perform two walking session per week, each consisting of 15*2-min walking bouts, with 2-min of rest in between. The intensity will be set at heart rate corresponding to the pain threshold.
  Arms: Walking training group

SUMMARY:
Whereas the efficacy of exercise interventions has been abundantly proven in male with peripheral artery disease (PAD), it remains to be determined whether these interventions are effective in women. The aim of this randomized controlled trial which will be performed with 34 PAD women will be to investigating the effects of 12 weeks of supervised walking on functional capacity and cardiovascular function and regulation at rest and during exercise.

ELIGIBILITY:
Inclusion Criteria:

* aankle-brachial index (ABI) ≤ 0.9 in one or two legs
* fontaine stage II of PAD
* body mass index <35 kg/m2
* resting systolic blood pressure (BP) <160 mmHg and diastolic BP <105 mmHg
* ability to walk at least 2min at 3.2 km/h
* ability to undertake an incremental treadmill test
* decrease of at least 15% in ABI after a maximal treadmill test
* not currently engaging in any regular exercise program

Exclusion Criteria:

* exercise induced signs of myocardial ischemia or complex ventricular arrhythmias
* cardiovascular autonomic neuropathy
* use of beta-blocker, nondihydropyridine calcium antagonists or insulin and hormone replacement therapy.

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Change in walking capacity at 12 weeks of follow-up | 12 weeks
  Claudication onset distance (m) defined as the distance walked until the patients first reported pain in the leg during the treadmill test and total walk distance (m) defined as the total distance that the patient was able to walk during the test will be performed before and after 12 weeks of follow-up.
Change in functional capacity at 12 weeks of follow-up | 12 weeks
  Walking economy defined as VO2 measured during the first stage of the treadmill test and functional capacity defined as VO2 peak obtained during the test will be measured to determine the cardiopulmonary response after 12 weeks of walking training.
Change in heart rate pain threshold at 12 weeks of follow-up | 12 weeks
  The heart rate obtained at claudication onset distance during the treadmill test will be evaluate before and after 12 weeks of follow-up.

SECONDARY OUTCOMES:
Change in Ankle-Brachial Index decrease at 12 weeks of follow-up | 12 weeks
  Will defined by the difference in ankle-brachial index measured immediately after the exercise and pre-exercise.
Change in ischemic window at 12 weeks of follow-up | 12 weeks
  Calculated by area under the curve of the ankle systolic blood pressure measured during the first 10 min of recovery after the test divided by total walk distance.
Change in autonomic modulation at 12 weeks of follow-up | 12 weeks
  Autonomic modulation: assessed by spectral analysis of heart rate and systolic blood pressure variabilities. Heart rate (electrocardiogram) and beat-by-beat blood pressure (finometer) will be recorded for 10 min at a sample frequency of 500Hz/channel.
Change in cardiac output at 12 weeks of follow-up | 12 weeks
  Cardiac output will be estimated at baseline and after 12 weeks of follow-up bu the indirect Fick method using the CO2 rebreathing technique and a metabolic card.
Change in vascular function at 12 weeks of follow-up | 12 weeks
  Blood flow and blood flow in response to hyperemia will be obtained.